CLINICAL TRIAL: NCT03818477
Title: Evaluation of TaqMan Array Card for Environmental Surveillance of Polio Virus and Antimicrobial Resistance Genes
Brief Title: Environmental Surveillance (ES) for Polio and AMR Using the TaqMan Array Card
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: University of Virginia (Other)
Collaborators: Bill and Melinda Gates Foundation (Other); International Centre for Diarrhoeal Disease Research, Bangladesh (Other)
Responsible Party: Principal Investigator, Mami Taniuchi, PhD, Assistant Professor, University of Virginia
Other Study IDs: 21092; PR-18038 (Other: International Centre for Diarrhoeal Disease Research)
Record Dates: First submitted 2019-01-24; First posted 2019-01-28 (Actual); Last update posted 2019-10-03 (Actual); Status verified 2019-10

CONDITIONS: Polio
MeSH Terms: conditions — Poliomyelitis

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study will be used to develop a tool to streamline poliovirus environmental surveillance for the polio endgame and to provide a tool for detecting polio in places where there is no capacity to carry out the gold standard culture-based detection.

DETAILED DESCRIPTION:
This environmental surveillance tool will also include antimicrobial resistance (AMR) genes to describe resistome profile in environmental samples and to better inform us of the potential risks of exposure to these environments

ELIGIBILITY:
Inclusion Criteria

* birth-4 years of age
* reside in selected urban slums of Mirpur Dhaka, Bangladesh
* receiving bOPV immunization

Exclusion Criteria:

* parent unwilling to consent

Max Age: 4 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The investigators will conduct a Supplementary Immunization Activity (SIA) using bivalent oral polio vaccine (bOPV) and administer bOPV to at least 70% of all children under the age of 5 in the participating wards in the urban slums of Mirpur, Dhaka
Sampling Method: Probability Sample
Enrollment: 8500 (Estimated)
Dates: Start 2019-06-09 (Actual); Primary Completion 2020-02-28 (Estimated); Study Completion 2020-09 (Estimated)

PRIMARY OUTCOMES:
Polymerase Chain Reaction (PCR) detection of poliovirus, enteric pathogens and antimicrobial resistance genes from environmental samples | through study completion, an average of 1 year
  Evaluate performance of the TaqMan Array Card (TAC) on environmental samples (sewage samples) collected in urban slum area of Mirpur. The primary purpose will be to use TAC to detect and monitor Sabin 1 and 3 polio viruses post SIA.

CONTACTS AND LOCATIONS:
Overall Officials: Mami Taniuchi, Principal Investigator — University of Virginia
Locations (1):
- International Centre for Diarrhoeal Disease Research, Dhaka, Bangladesh

IPD SHARING:
Plan to Share IPD: No